CLINICAL TRIAL: NCT06320106
Title: Evaluation of Spatial Navigation Skills in Typically Developing Children and in Children With Cerebral Palsy Using a Head Mounted Display
Brief Title: Assessment of Navigation Abilities in Children With Cerebral Palsy and Their Peers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GIP 1021
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Palsy; Healthy Volunteers
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CP group (Experimental): Participants with cerebral palsy are recruited.
  Interventions: Other: Virtual Reality baseline assessment
- TD group (Experimental): Typically developing children are recruited.
  Interventions: Other: Virtual Reality baseline assessment

INTERVENTIONS:
Other: Virtual Reality baseline assessment — They undergo a baseline assessment (including cognitive level and pen and paper tests for visuo-spatial abilities). Then they perform a spatial navigation assessment with an immersive virtual reality application delivered by the Oculus Quest viewer. The spatial navigation application consists of a 5-way star-maze adapted from (Biffi et al 2020 Front. Psychol.) where the participants have to find a treasure hidden at the end of one way. The application measures both the learning of spatial information and the strategy used (egocentric or allocentric).
  After the session, the participants fill questionnaires related to cyber-sickness and usability of the application.

SUMMARY:
Spatial navigation skills are very important in everyday activities and quality of life but spatial navigation abilities are not part of the standard process of assessment and rehabilitation of patients. Furthermore, it is known that children with cerebral palsy have impaired visuo-spatial competences. The main objective of this study is to evaluate and compare the spatial navigation abilities of typically developing children and of children with cerebral palsy using the "StarMaze" application delivered by means of a Head Mounted Display (HMD). The second aim is to investigate the user experience during the session. A similar application was already developed and tested in a virtual reality large scale platform whose size and cost limit the accessibility. Therefore, the assessment (and future training) of navigation abilities with affordable and easy-to-use technology such as HMD open new perspectives.

ELIGIBILITY:
Inclusion Criteria:

* IQ higher than 70

Exclusion Criteria:

* Subjects with epileptic issues
* Subjects with poor head control
* Visual acuity not correctable with eyeglasses

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Navigation strategy | One day
  The navigation strategy is measured by the application "StarMaze" delivered by the Oculus Quest viewer and it could be egocentric or allocentric. The strategy is egocentric if the participant finds the treasure in the virtual space by using a self-centred trajectory. The strategy is allocentric if the participant find the treasure in the virtual space by using a trajectory based on environmental cues.

SECONDARY OUTCOMES:
Learning rate | One day
  The learning rate of correct path to follow to find the treasure strategy is measured by the application "StarMaze" delivered by the Oculus Quest viewer. It is the number of trials required by the participant to reach a stable performance
Simulator Sickness Questionnaire | One day
  The questionnaire evaluates the effects of cyber sickness. Participants have to score 16 symptoms on a four-point scale (0-3).The symptoms can be placed into three general categories: oculomotor, disorientation, and nausea. Weights are assigned to each of the categories and summed together to obtain a single score.
System Usability Scale | One day
  It evaluates the usability of the system. The SUS is a simple, ten-item five-point Likert scale giving a global view of subjective assessments of usability.
Independent Television Commission-Sense of Presence Inventory | One day
  It is a 5-point Likert scale, composed of 44 items. This questionnaire evaluates the user experience to understand if the person enjoyed the game, the setting, and the overall experience. In particular, the questionnaire addresses four factors: spatial presence, engagement, realness of the environment, and side effects (cyber sickness).
Suitability Evaluation Questionnaire - simplified version | One day
  It evaluates the sense of agency with four questions (likert scale 1-5) and one open question.
Short-form of PANAS-Positive Affect and Negative Affect Scales | One day
  In the questionnaire, the participant must evaluate how much s/he feels in the way described by the adjective when filling out the questionnaire, responding on a 5-point Likert scale. The PANAS provides measures of Positive Affects (PAs) and Negative Affects (NAs). The PA and NA scores are the sums of the ratings of the PA items and the NA items, respectively. PA indicates the level of pleasurable engagement with the product while NA is a general factor of subjective distress.

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific Institute, IRCCS E. Medea, Bosisio Parini, Lecco, Italy